CLINICAL TRIAL: NCT04730206
Title: The DAWN Antivirals Trial: the Efficacy of Antivirals for COVID-19 Infections Presenting to Ambulatory Care: a Randomized Controlled Trial
Brief Title: The DAWN Antivirals Trial for Ambulatory COVID-19 Patients
Acronym: DAWN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment was too slow
Sponsor: KU Leuven (Other)
Collaborators: Universiteit Antwerpen (Other); University Ghent (Other); Université de Liège (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Ann Van den Bruel, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S64445
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — camostat; molnupiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be masked for camostat or placebo, molnupiravir is open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Camostat (Experimental): 4 x 200 milligram per day for 7 days
  Interventions: Drug: Camostat
- Placebo (Placebo Comparator): 4 x per day for 7 days
  Interventions: Drug: Placebo
- Molnupiravir (Experimental): 2 x 800 milligram per day for 5 days
  Interventions: Drug: Molnupiravir

INTERVENTIONS:
Drug: Camostat — 100 milligram tablets
  Arms: Camostat
Drug: Placebo — oral tablets, identical in size and shape
  Arms: Placebo
Drug: Molnupiravir — 200 milligram tablets
  Arms: Molnupiravir

SUMMARY:
This is a prospective, placebo controlled, individually randomized controlled phase III trial in Primary Care, assessing the efficacy of antivirals, i.e. camostat and molnupiravir, in accelerating recovery in Covid-19 patients.

DETAILED DESCRIPTION:
In patients aged 40 years and above and diagnosed with Covid-19 upon study entry, we will evaluate the efficacy of camostat or molnupiravir on recovery within 30 days after randomisation. Participants will be randomly assigned to camostat, molnupiravir or placebo using a computer generated randomisation process. Participants will be treated for 7 days in case of camostat and 5 days in case of molnupiravir, and follow-up will be 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older;
* At least 2 Covid-19 suggestive symptoms at the time of inclusion, with onset of a maximum of 5 days prior to enrolment, and which cannot be explained by an alternative cause, and defined by the current Sciensano case definition
* Positive result on PCR test or rapid Ag test in the 7 days before inclusion or at the time of inclusion;
* Patient is community dwelling;
* Participant or their proxy is willing and able to give informed consent for participation in the trial;
* Participant is willing to comply with all trial procedures.

Exclusion Criteria:

* Hospital admission is required at the time of possible recruitment;
* Positive PCR or rapid antigen test for SARS-CoV-2 in the last 2 months other than a test at recruitment or in the 7 days prior to recruitment;
* Participating in any other interventional drug clinical study before enrolment in the study;
* Breastfeeding;
* Known severe neurological disorder, especially seizures in the last 12 months;
* Known allergy to camostat or molnupiravir;
* Previous adverse reaction to, or currently taking, camostat or molnupiravir;
* Patients in palliative care;
* Pregnant women or women of childbearing potential who may become pregnant during the trial and don't agree to use any of the effective contraceptive measures lised above;
* Judgement of the recruiting clinician deems participant ineligible.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Time to first self-reported recovery within 30 days after randomisation | within 30 days after randomisation

SECONDARY OUTCOMES:
All-cause unplanned hospital admission for at least 24 hours | within 30 days after randomisation
All-cause mortality | within 30 days after randomisation
Health status | at 8 days and 30 days after randomization
  Score on the World Health Organisation (WHO) clinical progression scale: measure of illness severity across a range from 0 (not infected) to 10 (dead) where lower scores indicate a better outcome.
Oxygen administration in the home setting | over a period of 30 days after randomization
  Number of patients who had oxygen at least once
All-cause mortality at 1 year after randomization | at 1 year
Cardiovascular and thromboembolic complications | within 7 days and 30 days after randomization
  Number of events
Symptom duration for each individual symptom | over a period of 30 days after randomization
  Duration of symptoms reported by the patient in the patient diary as being present since randomisation
Duration of hospital admission for those admitted to hospital | over a period of 30 days after randomization
  Length of stay
Health services usage | over a period of 30 days after randomization
  Number of contacts with general practitioners, out-of-hours services, emergency department visits, specialist assessments
Consumption of antibiotics | over a period of 30 days after randomisation
  Antibiotic consumption expressed in defined daily dose
Participants' quality of life | at 7 days and 30 days after randomization
  Euroqol EQ-5D-5L: The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems, where higher scores indicate a better outcome
Time to sustained recovery within 14 days | within 30 days after randomisation
  time from randomization to self-reported recovery within 14 days and remaining recovered until day 30 after randomisation.
At least once ventilated | over a period of 30 days after randomization
Admission to ICU | over a period of 30 days after randomization
All-cause unplanned hospital admission for at least 24 hours or all-cause mortality within 30 days of randomization | over a period of 30 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium